CLINICAL TRIAL: NCT00147082
Title: Leukocyte Migration and Differentiation in COPD Patients Compared to Healthy Smokers and Healthy Non-smoking Subjects.
Brief Title: Leukocyte Function in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 01-024
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Results first posted 2019-12-05 (Actual); Last update posted 2019-12-05 (Actual); Status verified 2019-12

CONDITIONS: COPD; Emphysema; Chronic Bronchitis
Keywords: chemokine; chemokine receptor; neutrophil; lymphocyte; monocyte
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COPD: Patients with COPD - no intervention
- Smokers without COPD: Smokers without COPD - no intervention
- Non-smokers: Non-smokers with no history of respiratory disease - no intervention

SUMMARY:
The aim of this study is to investigate the mechanisms whereby leukocytes are recruited to the lung in chronic obstructive pulmonary disease (COPD) and cause tissue destruction. The hypothesis is that in COPD more leukocytes enter the lung and it is these cells that are responsible for the degradation of lung tissue. We, the researchers at Imperial College London, will isolate leukocytes from the blood of patients with COPD, healthy smokers and normal subjects and measure the movement of the leukocytes to chemoattractants. We will examine further, which cell surface receptors are responsible for this trafficking of cells. Furthermore, the differentiation of these cells in vitro will be compared with cells from healthy smokers and normal subjects. Specifically, the expression of enzymes that are responsible for tissue destruction and the cell surface receptors on these cells will be investigated. The objective is to identify the mechanisms whereby leukocytes from COPD patients behave differently to cells from healthy smokers and normal subjects with a view to identify novel targets for drug therapy.

DETAILED DESCRIPTION:
Chemotaxis experiments will be performed in order to ascertain the migratory characteristics of leukocytes towards specific chemoattractants. Comparisons of cells from different subjects will be compared. In addition, the effects of various pharmaceutical interventions on this mechanism will also be addressed and compared within subject groups. In some experiments, cells will be differentiated in vitro and their cellular expression and regulation of inflammatory mediators and chemoattractants examined. Again comparisons will be made between subject groups and the efficacy of various pharmacological agents on these cells

ELIGIBILITY:
Inclusion Criteria:

* Healthy Non-Smoking Subjects. All normal volunteers will meet the following criteria:

  * Age 21-70 years.
  * No history of respiratory or allergic disease.
  * Normal baseline spirometry as predicted for age, sex and height.
  * Non-smokers.
  * No history of upper respiratory tract infection in the preceding six weeks.
  * Not taking regular medication
* COPD Subjects. COPD is diagnosed according to American Thoracic Society, European Respiratory Society and British Thoracic Society guidelines. All COPD volunteers will meet the following criteria:

  * Age between 40-75 years.
  * A smoking history of at least 20 pack years. (1 pack year = 20 packs of cigarettes per day for 1 year)
  * Forced expiratory volume at 1 second : Forced vital capacity (FEV1:FVC) ratio of <0.7, post-bronchodilator FEV1 of <85% predicted, reversibility with inhaled beta2-agonist of <15% of predicted FEV1: all three criteria are required.
  * Current smokers or smokers who had ceased smoking for at least 6 months.
  * No history of exacerbation, oral steroid or antibiotic use within the preceding 6 weeks.
  * Normal serum alpha-1 antitrypsin level.
  * No history of other respiratory or allergic disease.
  * No evidence of atopy on skin prick testing to common aeroallergens (grass pollen, cat hair, house dust mite or Aspergillus fumigatus
* Healthy Smokers. All healthy smoking volunteers in trials will meet the following criteria:

  * Age 21-70 years.
  * Smoking history of at least 10 pack years. (1 pack year = 10 packs of cigarettes per day for 1 year).
  * No history of respiratory or allergic disease.
  * Normal baseline spirometry as predicted for age, sex and height.
  * No history of upper respiratory tract infection in the preceding six weeks.
  * Not taking regular medication.

Exclusion Criteria:

Subjects will not be included in this study if they meet any of the following exclusion criteria:

* Clinically significant findings in the medical history or on physical examination other than those of COPD in the COPD group.
* Pregnant women or mothers who are breastfeeding.
* Subjects who are unable to give informed consent.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who had taken inhaled or oral steroids or who had suffered an exacerbation of their airway disease in the previous 6 weeks were excluded.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2001-02 (Actual); Primary Completion 2004-12 (Actual); Study Completion 2007-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Louise E Donnelly, PhD, Principal Investigator — Imperial College London
Locations (1):
- Royal Brompton Hospital/NHLI Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Traves SL, Smith SJ, Barnes PJ, Donnelly LE. Specific CXC but not CC chemokines cause elevated monocyte migration in COPD: a role for CXCR2. J Leukoc Biol. 2004 Aug;76(2):441-50. doi: 10.1189/jlb.1003495. Epub 2004 May 20. PMID 15155777

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | COPD | Smokers Without COPD | Non-smokers
Started | 37 | 33 | 30
Completed | 37 | 33 | 30
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | COPD | Smokers Without COPD | Non-smokers | Total
Number analyzed (Participants) | 37 | 33 | 30 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 65 (10) | 40 (12) | 34 (8) | 47.45 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 15 | 13 | 41
  Male | 24 | 18 | 17 | 59
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 37 | 33 | 30 | 100
Smoking History [Mean (Standard Deviation); unit: pack/years] | 48 (27) | 21 (16) | 0 (0) | 24.7 (21)
FEV1 (% predicted) [Mean (Standard Deviation); unit: % predicted] | 47 (15) | 93 (21) | 102 (14) | 78.7 (17)

OUTCOME MEASURES:

1. Primary Outcome: Effective Concentration (EC 50) of GRO Alpha
Description: Migration response of PBMC to Chemokine EC 50 represents the concentration of a drug that is required for 50% inhibition in vitro
Time Frame: 2 hours
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | COPD | Smokers Without COPD | Non-smokers
Number analyzed (Participants) | 37 | 33 | 30
ng/ml | 1.5 (0.9) | 0.9 (0.2) | 0.6 (0.3)
Statistical Analysis 1: Comparison: COPD vs Smokers Without COPD vs Non-smokers; p values were calculated; Test type: Superiority; p = 0.05, Kruskal-Wallis — The threshold for significance was p<0.05

2. Primary Outcome: Effective Concentration of IL-8
Description: as for outcome 1
Time Frame: 2 hours
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | COPD | Smokers Without COPD | Non-smokers
Number analyzed (Participants) | 37 | 33 | 30
ng/ml | 0.2 (0.1) | 1.4 (0.4) | 0.8 (0.4)
Statistical Analysis 1: Comparison: COPD vs Smokers Without COPD vs Non-smokers; p value was calculated; Test type: Superiority; p = 0.05, Kruskal-Wallis — The p value (<0.05) was the threshold for significance

3. Primary Outcome: Effective Concentration of MCP-1
Description: Migration response of PBMC to Chemokine
Time Frame: 2 hours
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | COPD | Smokers Without COPD | Non-smokers
Number analyzed (Participants) | 37 | 33 | 30
ng/ml | 0.5 (0.4) | 0.2 (0.2) | 0.3 (0.3)
Statistical Analysis 1: Comparison: COPD vs Smokers Without COPD vs Non-smokers; The p value was calculated; Test type: Superiority; p = 0.05, Kruskal-Wallis — The p value (<0.05) was the threshold for significance

ADVERSE EVENTS:
Time Frame: 2 hours
Arm/Group | COPD | Smokers Without COPD | Non-smokers
All-Cause Mortality (participants affected / at risk) | 0/37 | 0/33 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/37 | 0/33 | 0/30
Other Adverse Events (participants affected / at risk) | 0/37 | 0/33 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes